CLINICAL TRIAL: NCT04352387
Title: Effects of a Culturally Adapted Group Based Montessori Based Activities on Engagement and Affect in Chinese Older People With Dementia
Brief Title: Montessori Based Activities for Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Food and Health Bureau, Hong Kong (Other Government)
Collaborators: The Salvation Army, Hong Kong and Macau Command (Other)
Responsible Party: Principal Investigator, Dr. Helen YL Chan, Associate Professor, Food and Health Bureau, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SA2019
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Dementia
Keywords: person-centered; community support
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two research assistants who conducted the observations were blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Montessori Method for Dementia (Experimental): The design of the Montessori Method for Dementia program covered five aspects, namely cognitive stimulation, life skills, motor movements and fitness, sensory stimulation, and socialization. Each 1-hour session included two to three activities tailored to the local cultural context.
  Interventions: Behavioral: Montessori Method for Dementia
- Usual care (Active Comparator): Activities delivered regularly in the usual care, such as reading out newspapers, physical activities, and watching videos, in the 1-hour sessions.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Montessori Method for Dementia — The Montessori Method highlights the importance of considering the past experiences, identifying interests and maximizing spared capacity and abilities of each individual.
  Arms: Montessori Method for Dementia
Behavioral: Usual care — Activities delivered regularly in the usual care, such as reading out newspapers, physical activities, and watching videos, in the 1-hour sessions.
  Arms: Usual care

SUMMARY:
The objectives of this study are to examine the feasibility of a culturally-adapted group-based Montessori Method for Dementia program in Chinese community and examine its effects on engagement and affect in community-dwelling people with dementia.

DETAILED DESCRIPTION:
People who were aged 60 years or over and with mild to moderate dementia were recruited from six community centres and three care homes. Participants were randomly assigned to either the intervention group to attend the Montessori-based activities or the comparison group to attend the conventional group activities for one hour twice per week over eight weeks. All sessions were videotaped to facilitate analysis. Observations of engagement and affect were conducted for each intervention session on the individual participant for a ten-minute period at the beginning, middle, and end of the activity in order to have observations from multiple time points. The Menorah Park Engagement Scale and the Apparent Affect Rating Scale were used to assess the engagement and affect during the activities based on observations.

ELIGIBILITY:
Inclusion Criteria:

* with a diagnosis of dementia at a stage 3 to 5 on the global deterioration scale (GDS)

Exclusion Criteria:

* were joining any other dementia training activities
* would highly likely present a hazard to others through disruptive behaviors
* proxy consent could not be obtained

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Engagement between the 1st minute - 10th minute of each session | through study completion for 8 weeks
  Score of Menorah Park Engagement Scale will be used to assess the level of engagement, with the minimum score of 0 and the maximum of 2, with a higher score higher level of engagement.
Engagement between the 25th minute - 35th minute of each session | through study completion for 8 weeks
  Score of Menorah Park Engagement Scale will be used to assess the level of engagement, with the minimum score of 0 and the maximum of 2, with a higher score higher level of engagement.
Engagement between the 50th minute - 60th minute of each session | through study completion for 8 weeks
  Score of Menorah Park Engagement Scale will be used to assess the level of engagement, with the minimum score of 0 and the maximum of 2, with a higher score higher level of engagement.
Affect between the 1st minute - 10th minute of each session | through study completion for 8 weeks
  Score of the Apparent Affect Rating Scale will be used to assess the level of affect, with 1 (Never) to 5 (over 5 minutes), in the aspect of pleasure and interest.
Affect between the 25th minute - 35th minute of each session | through study completion for 8 weeks
  Score of the Apparent Affect Rating Scale will be used to assess the level of affect, with 1 (Never) to 5 (over 5 minutes), in the aspect of pleasure and interest.
Affect between the 50th minute - 60th minute of each session | through study completion for 8 weeks
  Score of the Apparent Affect Rating Scale will be used to assess the level of affect, with 1 (Never) to 5 (over 5 minutes), in the aspect of pleasure and interest.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Chan, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Salvation Army, Hong Kong and Macau Command, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan HY, Yau YM, Li SF, Kwong KS, Chong YY, Lee IF, Yu DS. Effects of a culturally adapted group based Montessori based activities on engagement and affect in Chinese older people with dementia: a randomized controlled trial. BMC Geriatr. 2021 Jan 7;21(1):24. doi: 10.1186/s12877-020-01967-0. PMID 33413153